CLINICAL TRIAL: NCT05225792
Title: Improved Training Method for Advanced Rehabilitation of Warfighters With Lower Extremity Trauma
Brief Title: Rapid Rehabilitation to Treat Lower Extremity Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenton R. Kaufman, PhD, PE, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-010009
Record Dates: First submitted 2021-12-08; First posted 2022-02-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Lower Limb Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injured Service Members (Experimental)
  Interventions: Behavioral: Promis Physical Function Questionnaire; Behavioral: L Test; Behavioral: Narrowing Beam Walking Test; Behavioral: PEQ-A

INTERVENTIONS:
Behavioral: Promis Physical Function Questionnaire — Patient reported physical function outcomes
Behavioral: L Test — Performance based measure assessing general physical function and balance ability.
Behavioral: Narrowing Beam Walking Test — Subjects attempt to walk along 4 progressively narrower beam segments with their arms crossed over their chest.
Behavioral: PEQ-A — Survey on confidence, stumbles and falls.
  Other Names: Prosthesis Evaluation Questionnaire - Addendum

SUMMARY:
The purpose of this study is to find out if an advance balance perturbation training program can enhance the rehabilitation process by increasing weight-bearing strategies on the prosthetic or injured limb, and, help reduce stumbles and falls.

ELIGIBILITY:
Inclusion Criteria:

* Research participants will be eligible active duty service members and retired veterans.
* Having lower limb trauma (transtibial and transfemoral amputations, bilateral amputations, and limb salvage).
* Are enrolled in conventional rehabilitation at the participating military treatment centers.
* Subjects with dysvascular disease will be excluded because compromised lower limb somatosensation and circulation are independently linked with poor postural stability and a history of frequent falls.
* For subjects with amputations, the individual must be a community ambulator (i.e., K-Level 3 or 4).
* For subjects with limb salvage, they will need to have an IDEO and be entered into the Return-to-Run training program.

Exclusion Criteria:

- Subjects must not have excessive pain or other neuromuscular problems that preclude them from performing the test protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prosthesis Evaluation Questionnaire-Addendum (PEQ-A) | 0, 6 months
  Fall incidence change between baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenton Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States